CLINICAL TRIAL: NCT04773821
Title: Performance of Prostate MRI and Targeted Biopsy to Detect Residual Prostate Cancer Following Focal Therapy
Brief Title: Performance of Prostate MRI and Following Biopsy to Detect Prostate Cancer Recurrence After Focal Therapy
Acronym: IRMProft
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP191126; 2020-A01466-33 (Other: IDRCB)
Record Dates: First submitted 2021-02-15; First posted 2021-02-26 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2021-09

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Focal Therapy; Multiparametric MRI; Prostate Specific Antigen; Prostate Specific Antigen density; Standard Biopsy; Targeted Biopsy; Trans rectal ultrasound; Trans rectal ultrasound guided biopsy; Non targeted Biopsy (Standard biopsy and zonal ablation); Cryotherapy; High-intensity focused ultrasound (HIFU); Irreversible electroporation; Laser ablation therapy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Arm (Experimental): All men patients with low and intermediate risk prostate cancer (ISUP 1 and 2) who has already chosen to undergo focal treatment, in the referral centers and responding to the inclusion criteria will be included after obtaining their writing consent. Follow-up visits are planned at 3, 6,12 and 13 month from the date of the focal treatment consistently with usual care. All patients will have a MpMRI and MpMRI targeted biopsy in the presence of a lesion suggestive of recurrence at 12 months. The subject will be his own control
  Interventions: Other: Targeted biopsies

INTERVENTIONS:
Other: Targeted biopsies — Prostate MpMRI at 12 month (after PCa focal treatment in standard care) and targeted biopsies in the presence of lesion(s) suggestive(s) of recurrence

SUMMARY:
The management of localized prostate cancer remains controversial because of a risk of over diagnosis and over treatment. Focal therapy represents an approach to improve the therapeutic ratio of prostate cancer treatments. Focal therapy has been developed as minimally invasive procedure with the aim of providing equivalent oncological safety, reduced toxicity and improved functional outcomes. Multiparametric (mp) MRI Imaging may provide a reliable mean of monitoring for disease recurrence, and has been suggested as the most accurate imaging tool currently available for systematic detection of recurrence, pre-biopsy and preoperative mapping for an eventual salvage therapy. However, question about the performance of MRI and targeted biopsy in monitoring and defining successful therapy and follow up has been poorly evaluated. Modalities (standard biopsy, ablation zone biopsy vs targeted biopsy) and number of biopsies to be performed, depending on the results of MRI, remains unanswered due to a lack of available data.

We hypothesize that the combination of MpMRI of the prostate with subsequent targeted biopsy (TB) may improve detection of prostate cancer and may therefore improve the follow-up of men after focal therapy (FT) to better identify patients that need a salvage treatment and when.

DETAILED DESCRIPTION:
This trial is a multi-centric prospective and diagnostic study, comparative, not randomised. The main objective is to evaluate the value of Multiparametric MRI (MpMRI) and targeted biopsy in detecting recurrence after focal treatment of prostate cancer (PCa). The secondary objectives (all energy and according to the energy used) are: to describe the specific changes in prostate morphology after focal therapy ( normal presentation and recurrence in the treated and in the non-treated zone, all energy and according to the energy used),to evaluate the accuracy of MpMRI in the detection of residual PCa, in the treated zone, in the whole gland, to evaluate the performance of targeted biopsy and non targeted biopsy for the detection of prostate cancer recurrence, to evaluate the combination of targeted biopsy and non targeted biopsy for the detection of prostate cancer recurrence, to assess the number and amount of unnecessary non targeted biopsies taken during the follow up of men in focal therapy, to describe the morbidity of prostate non-targeted and targeted biopsy (number and severity of biopsy complications) for the detection of prostate cancer recurrence, to evaluate the impact of recurrence detection on patient management (number and type of salvage treatment),to evaluate the post treatment PSA levels including density, PSA nadir, and its goal in detection recurrence, to examine failures in order to learn potential future predictors of failure (all energy and according to the energy used, the initial location of the target on MRI and it's Gleason grade).The first objective of ancillary study is a central MRI lecture with 3 experts which will allow, performance and inter-observer reproducibility, to evaluate the percentage of cases that will be scored with agreement for concordant biopsy decision by the central radiology team and the site radiologist, to determine on the pre-treatment MRI predictive criteria of success or failure for focal therapy according of the energy used and to propose recommendations for MRI interpretation after FT. The second objective of ancillary study is a central pathology reading to evaluate the percentage of cases that will be scored with agreement on the Gleason score by the central pathologists and the site pathologist and to propose recommendations for histology interpretation post focal therapy. The study population will consist of men with low and intermediate risk prostate cancer (ISUP 1 and 2) who has already chosen to undergo focal treatment, and be willing and able to undergo MpMRI with subsequent prostate biopsies, as indicated. Patients will be enrolled at baseline by an urologist in one of urology units listed as investigation center. The focal treatment should take place no later than 3 months after inclusion visit. The follow-up visits will be planned at 3 month,6 month,12 and 13 months after focal treatment, consistently with patient usual care. In this study, all patients will have a MpMRI and MpMRI targeted biopsy in the presence of a lesion suggestive of recurrence.The statistical analysis is to compare the positive biopsy rate between non targeted and targeted in subject as his own control (with a 12-month relapse rate of 30%) assuming 18.25% positive with the standard method (H0) and 26.25% with the targeted method (H1) and 15% of discordant pairs. By simulation with a MacNemar test, with a bilateral alpha risk of 5% and power of 90% we need 260 subjects.

ELIGIBILITY:
Inclusion criteria

1. Age > 18 years
2. Detection of prostate cancer must have be done by combination of MRI plus biopsy following (EAU guidelines and French Guidelines)
3. Patient had no prior treatment for PCa
4. The patient could be classified as low- or intermediate-risk, according to D'Amico's 2003 [15] risk group categories: T1c, T2a, PSA less than 20ng/ml, with Gleason Grade of 6 (3+3) or 7 (3+4 ) (ISUP 1 and ISUP 2)
5. Management decisions should be made after all treatments have been discussed in a multidisciplinary team and after the balance of benefits and side-effects of appropriate therapy modalities has been considered together with the patient.
6. Patient informed of treatment options and have already chosen to undergo focal treatment (focal, quadrant or hemi-ablation) by cryotherapy, high-intensity focused ultrasound (HIFU), irreversible electroporation, laser ablation therapy (including photodynamic therapy) and microwave
7. Preoperative MRI and biopsy results will be mandatory
8. Participant must be willing to attend the follow up visits
9. Participant must be willing and able to attend follow-up MRI and prostate biopsies
10. Written informed consent
11. Affiliation to a French social security system excluding AME (Aide médicale d'état)

Exclusion criteria

1. Hormone therapy within the past year
2. Prior pelvic radiotherapy
3. Focal brachytherapy
4. Concurrent participation in other interventional clinical studies with radical treatment of prostate cancer
5. Contraindications to undergo MpMRI or Trans rectal ultrasound TRUS-guided prostate biopsy (TRUS-Bx)
6. Patient deprived of liberty or under legal protection measure

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2021-06-02 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
The detection rate of prostate cancer after focal treatment | At 12 months after focal treatment
  To compare the detection rates obtained by both standard (STB) and targeted methods (TB), both types of biopsy being done on the same subjects

SECONDARY OUTCOMES:
PCa detection on the combination of Targeted Biopsy (TB) and Non targeted Biopsy (NTB) | At 12 months after focal treatment
  To estimate the detection of Pca by the combination of the TB and NTB at once, and determinate the sensibility and the specificity in this configuration of combination.
Morbidity of prostate biopsy | through the study completion, an average of 40 months
  Nature and severity of short term and long term biopsy complications: infection, hemorrhage, other
Number of salvage treatment by focal therapy | through the study completion, an average of 40 months
Number of salvage treatment by radical prostatectomy | through the study completion, an average of 40 months
Number of salvage treatment by external radiotherapy | through the study completion, an average of 40 months
Prostate Specific Antigen (PSA) | at 3 months, 6 months,12 months
Prostate Specific Antigen density (PSAd) | at 3 months and 12 months
Accuracy of MpMRI to detect PCa after focal treatment | At 12 month after focal treatment
Number of positive MpMRI | through the study completion, an average of 40 months
  Number of positive MpMRI define by a Likert score > =3 in the treated and the non-treated zone
Localization of positive MpMRI | through the study completion, an average of 40 months
  Localization of positive Mp MRI define by a Likert score > =3 in the treated and the non-treated zone

CONTACTS AND LOCATIONS:
Overall Officials: Raphaële RENARD PENNA, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (11):
- France (11):
  - CHRU Brest - Hôpital de la Cavale Blanche, Brest
  - CH Chartres - Hôpital Louis Pasteur, Chartres
  - CHU DIJON Francois Mitterrand, Dijon
  - CHU de Nice Hôpital Pasteur 2, Nice
  - Groupe Hospitalier Pitié Salpêtrière, Paris
  - Hôpital Tenon, Paris
  - Hôpital Cochin, Paris
  - Institut Mutualiste Montsouris, Paris
  - Clinique La Croix du Sud Quint-Fonsegrives, Quint-Fonsegrives
  - CHU de Rennes - Hôpital Pontchaillou, Rennes
  - Hôpital Foch, Suresnes

IPD SHARING:
Plan to Share IPD: No